CLINICAL TRIAL: NCT03843086
Title: Safety and Efficacy of Low Intensity Shockwaves for the Treatment of Erectile Dysfunction - Comparison of Two Treatment Schedules
Brief Title: Low Intensity Linear Shockwave Therapy for Erectile Dysfunction
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in device and protocol
Sponsor: University of Virginia (Other)
Collaborators: DIREX SYSTEMS CORPORATION (Industry)
Responsible Party: Principal Investigator, Ryan Smith, MD, Assistant Professor of Urology, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21221
Record Dates: First submitted 2019-01-28; First posted 2019-02-15 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Vasculogenic Erectile Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 720 Low Intensity shockwave therapy (Active Comparator): Five daily sessions within a week, Monday thru Friday, in which 720 shocks of treatment energy applied every session to each treated region (left and right corpora cavernosa and crura)
  Interventions: Device: Low Intensity Linear Shockwave Device for the treatment of Erectile Dysfunction
- 600 Low Intensity shockwaves therapy (Active Comparator): Three weekly sessions for 2 consecutive weeks, Monday-Wednesday-Friday, in which 600 shocks of treatment energy applied every session to each treated region (left and right corpora cavernosa and crura)
  Following the last treatment session, each patient will resume his baseline consumption of phosphodiesterase 5 inhibitor in terms of type and dose of drug, for the remainder of study duration.
  Interventions: Device: Low Intensity Linear Shockwave Device for the treatment of Erectile Dysfunction

INTERVENTIONS:
Device: Low Intensity Linear Shockwave Device for the treatment of Erectile Dysfunction — This is a prospective, randomized, clinical study aimed to evaluate the safety and efficacy of the two treatment schedules on symptomatic erectile dysfunction patients using low intensity shockwave therapy. The patients are randomized in a 1:1 ratio into two active treatment groups.
  Group A: 5 daily sessions within a week (Monday, Tuesday, Wednesday, Thursday, Friday), in which 720 shocks of treatment energy will be applied in every session to each treated region (left and right corpora cavernosa and crura).
  Group B: Three sessions per week (Monday, Wednesday, Friday) for 2 consecutive weeks, in which 600 shocks of treatment energy will be applied in every session to each treated region (left and right corpora cavernosa and crura)
  Other Names: MoreNova

SUMMARY:
MoreNovaED is a Linear Shockwaves (LISW) device in which shockwaves are focused onto line segments for improved organ coverage. Shockwaves produced by MoreNovaED are aimed at the left and right corpora cavernosa and the crura. The study is aimed at determining the safety and effectiveness of this new type LISW in the relief of ED.

DETAILED DESCRIPTION:
Morenova-Erectile dysfunction (ED) is a Linear Shockwaves (LISW) device which incorporates a unique shockwave transducer operable to deliver shockwaves to a treated region confined to a narrow rectangle. Shockwaves generation follows the electromagnetic principle. Low intensity shockwaves do not inflict pain and anesthesia or sedation is not required.

This current study is a prospective, pilot, randomized, uncontrolled clinical study aimed to evaluate the safety and efficacy of the two treatment schedules on symptomatic ED patients. The patients are randomized in a 1:1 ratio into active treatment groups.

Rationale:Linear Shockwaves has been known to bolster angiogenesis by increasing the levels of vascular endothelial growth factor.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has been correctly informed about the study
2. The patient must have given his informed and signed consent
3. The patient is a man between 40 and 80 years of age
4. The patient has ED of Vasculogenic origin
5. The patient is PDE5i responsive, meaning he is able to achieve and maintain an erection under the effect of the maximal dosage of PDE5i
6. The patient has been in a stable heterosexual relationship for over 3 months prior to enrollment
7. A minimum of 2 sexual attempts per month for at least one month prior to enrollment
8. The patient is suffering from erectile dysfunction lasting for over 6 months and not more than 5 years
9. IIEF-EF score between 17 and 25
10. Testosterone level 300-1000 ng/dL within 1 month prior to enrollment
11. A1C level ≤ 7% within 1 month prior to enrollment
12. Patients have at least a natural tumescence during sexual stimulation (EHS score ≥ 1).

Exclusion Criteria:

1. The patient is participating in another study that may interfere with the results or conclusions of this study
2. Within the past three months, the patient has participated in another study that may interfere with the results or conclusions of this study
3. The patient is in an exclusion period determined by a previous study
4. The patient is under judicial protection
5. The patient is an adult under guardianship
6. The patient refuses to sign the consent
7. It is impossible to correctly inform the patient
8. History of radical prostatectomy or extensive pelvic surgery
9. Venous leak
10. Past radiation therapy of the pelvic region within 12 months prior to enrollment
11. Recovering from cancer within 12 months prior to enrollment
12. Neurological disease which effects erectile function
13. Psychiatric disease which effects erectile function
14. Anatomical malformation of the penis, including Peyronie's disease
15. Testosterone level <300 or >1000 ng/dL within 1 month prior to enrollment
16. A1C level > 7% within 1 month prior to enrollment
17. The patient is taking blood thinners and has an international normalized ratio >3.

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2019-06 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
International Index of Erectile Function (IIEF-EF) Questionnaire | 7 months
  The 15-question International Index of Erectile Function (IIEF) Questionnaire is a validated, multi-dimensional, self-administered investigation that has been found useful in the clinical assessment of erectile dysfunction and treatment outcomes in clinical trials

SECONDARY OUTCOMES:
SEP (Sexual Encounter Profile) 2 & 3 at follow-ups | 7 months
  Sexual activity improvement leading to optimal penetration at follow-ups. 2 Yes or No questions
GAQ (Global Assessment Questions) at follow-ups | 7 months
  2 Yes or No questions assessing improvement with treatment
EHS (Erection Hardness Score) at follow-ups | 7 months
  Scale rating hardness of erection from 0-4 with 4 being highest

CONTACTS AND LOCATIONS:
Overall Officials: Ryan P Smith, M.D., Principal Investigator — University of Virginia

IPD SHARING:
Plan to Share IPD: Undecided